CLINICAL TRIAL: NCT00871416
Title: Localisation of Potential Insulin Deposits in Normal Weight and Obese Diabetics Using 6 mm and 12 mm Long Needles. Furthermore, the Thickness of Cutis/Subcutis Is Measured on Recommended Insulin Injection Sites
Brief Title: Localisation of Potential Insulin Deposits in Normal Weight and Obese Diabetics Using 6 mm and 12 mm Long Needles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NEEDLEN/DCD/3/DK
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Delivery Systems
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: NovoFine® needle 6 mm
  Other Names: NEEDLEN
Device: NovoFine® needle 12 mm
  Other Names: NEEDLEN

SUMMARY:
This trial is conducted in Europe. The primary aim of this clinical trial is to locate and compare simulated insulin injections (injections of sterile atmospheric air) in normal weight and obese patients with diabetes mellitus. Injections are done with 6 mm and 12 mm needles with and without lifting of skin fold at different injection sites.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Use NovoPen®, NovoPen® 1.5, NovoPen® 3, NovoLet® 1.5 or NovoLet® 3 for at least 3 months
* Body mass index (BMI) for normal weight between 19-25 kg/m2
* Body mass index (BMI) for obese between 25-33 kg/m2

Exclusion Criteria:

* Pregnancy or plans thereof
* Local reactions on injection sites
* Acute, severe infection diseases
* Coagulation disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1997-04-09 (Actual); Primary Completion 1997-07-18 (Actual); Study Completion 1997-07-18 (Actual)

PRIMARY OUTCOMES:
Location of the injected sterile, atmospheric air | after 4 injections at visit 1 and 2, respectively

SECONDARY OUTCOMES:
Cutis/subcutis thickness on 14 recommended injection sites

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Aarhus, Denmark

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com